CLINICAL TRIAL: NCT02216942
Title: Endodontic Treatment of Primary Teeth With Guedes Pinto Paste: A Randomized Clinical Trial
Brief Title: Endodontic Treatment of Necrotic Primary Teeth With Guedes Pinto Paste: A Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fausto Medeiros Mendes (Other)
Responsible Party: Sponsor-Investigator, Fausto Medeiros Mendes, Fausto Medeiros Mendes, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOUSP2408
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Endodontic Treatment of Primary Teeth
Keywords: Endodontics; Deciduous teeth; Iodoform pastes; Treatment Refusal
MeSH Terms: conditions — Treatment Refusal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitapex (Active Comparator): Endodontic treatment using Vitapex
  Interventions: Drug: Endodontic treatment using Vitapex
- Guedes Pinto Paste (Experimental): Endodontic treatment using Guedes Pinto
  Interventions: Drug: Endodontic treatment using Guedes Pinto

INTERVENTIONS:
Drug: Endodontic treatment using Vitapex — Endodontic treatment using Vitapex
  Arms: Vitapex
Drug: Endodontic treatment using Guedes Pinto — Endodontic treatment using Guedes Pinto paste
  Arms: Guedes Pinto Paste

SUMMARY:
The maintenance of primary teeth until their exfoliation has been one of the main purposes of Pediatric Dentistry, are they representing the fundamental basis for proper occlusion of the permanent dentition. Often, injuries or extensive dental caries reach the pulp of deciduous teeth making maintenance on these dependent endodontic treatment arc. Thus, this study was to conduct a randomized clinical trial with longitudinal follow-up of two years, double blind, to compare the degree of success of endodontic treatment in primary among the most used folder, Guedes Pinto paste, and one Calcium hydroxide and iodoform paste to control, Vitapex.

DETAILED DESCRIPTION:
After approval by the ethics committee of the patients Faculty of Dentistry, University of São Paulo that having root canal filling of primary teeth will be invited to participate in the study. A clinical examination and prior radiographic diagnosis and also a quality of life questionnaire regarding oral health (- ECOHIS Early Childhood Oral Health Impact Scale) will be-held. The patient will be randomized to one of two groups and will be held endodontics by a blind handler. The patient will be accompanied with periods of one week, six months, 12 months and 24 months by a blinded evaluator. At the last visit of the review ECOHIS questionnaire will be reapplied to those responsible. The outcome will be the success or failure of endodontic treatments evaluated through permanent tooth in the arch on clinical and radiographic conditions of normality. The longevity of the treatments will be evaluated by estimating survival rates by Kaplan-Meier. The differences between the survival rates according to the type of proposed endodontic treatment will be analyzed using the log-rank test with a minimum significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Primary teeth with pulp diagnosis and need endodontic treatment
* Patients whose guardians consent to their participation in the survey
* fistula or abscess
* bone rarefaction or visual diagnosis
* teeth in the remaining tooth structure and location of the injury rehabilitation permit
* do not have internal or external resorption involving more than one third of the root length
* have no bone loss in lateral root and disruption crypt and the presence of at least half of root

Exclusion Criteria:

* health problems systemic
* congenital facial deformities
* facial tumors
* syndromes

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Success or failure of two endodontic treatments | two years
  The success or failure of endodontic treatments evaluated by the time spent in the tooth arch in clinical conditions of normality. Clinical criteria for determining success are: absence of fistula, absence of painful symptoms and pathological absence of adequate mobility and gingival contour. Radiographically, the success criteria are: absence / reduction of periapical bone rarefaction in anterior and absence / bone rarefaction in the furcation area of later, maintaining the periradicular space, root resorption compatible with the eruptive phase and absence of pathological bone resorption. To evaluate the reduction of lesions or appearance of new lesions will be between the initial and follow-up radiographs. Radiographs will be scanned and the end of the bone rarefactions starting area and will be measured on a software image analysis.

SECONDARY OUTCOMES:
Quality of the obturation obtained with the two root canal filling pastes | two years
  The quality of the filling will be assessed by a blinded examiner according to two criteria. Through an index that ranks the shutter in satisfactory, questionable or unsatisfactory and through evaluation of digital radiographic images with the aid of a computational tool (Autodesk AutoCAD), where the visible areas of the root canal will be measured in previous radiographic examination and their measurements of the area of the root canal filling pastes filled with channels. The influence of the quality of the filling in the successful treatment will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Bresolin, PHD student, Principal Investigator — University of Sao Paulo
Locations (1):
- Carmela Bresolin, São Paulo, Brazil

REFERENCES:
- [Background] Kopel HM. Root canal therapy for primary teeth. J Mich State Dent Assoc. 1970 Feb;52(2):28-33 passim. No abstract available. PMID 5263926
- [Background] Garcia-Godoy F. Evaluation of an iodoform paste in root canal therapy for infected primary teeth. ASDC J Dent Child. 1987 Jan-Feb;54(1):30-4. PMID 3468139
- [Background] Rifkin A. A simple, effective, safe technique for the root canal treatment of abscessed primary teeth. ASDC J Dent Child. 1980 Nov-Dec;47(6):435-41. No abstract available. PMID 6934178
- [Background] Rifkin A. The root canal treatment of abscessed primary teeth--a three to four year follow-up. ASDC J Dent Child. 1982 Nov-Dec;49(6):428-31. No abstract available. PMID 6960030
- [Background] Fuks AB. Pulp therapy for the primary and young permanent dentitions. Dent Clin North Am. 2000 Jul;44(3):571-96, vii. PMID 10925773
- [Background] Kubota K, Golden BE, Penugonda B. Root canal filling materials for primary teeth: a review of the literature. ASDC J Dent Child. 1992 May-Jun;59(3):225-7. PMID 1629445
- [Background] Mass E, Zilberman UL. Endodontic treatment of infected primary teeth, using Maisto's paste. ASDC J Dent Child. 1989 Mar-Apr;56(2):117-20. PMID 2656788
- [Background] Srinivasan V, Patchett CL, Waterhouse PJ. Is there life after Buckley's Formocresol? Part I -- a narrative review of alternative interventions and materials. Int J Paediatr Dent. 2006 Mar;16(2):117-27. doi: 10.1111/j.1365-263X.2006.00688.x. PMID 16430526
- [Background] Waterhouse PJ, Nunn JH, Whitworth JM, Soames JV. Primary molar pulp therapy--histological evaluation of failure. Int J Paediatr Dent. 2000 Dec;10(4):313-21. doi: 10.1046/j.1365-263x.2000.00211.x. PMID 11310245
- [Background] Wright KJ, Barbosa SV, Araki K, Spangberg LS. In vitro antimicrobial and cytotoxic effects of Kri 1 paste and zinc oxide-eugenol used in primary tooth pulpectomies. Pediatr Dent. 1994 Mar-Apr;16(2):102-6. PMID 8015949
- [Background] Mani SA, Chawla HS, Tewari A, Goyal A. Evaluation of calcium hydroxide and zinc oxide eugenol as root canal filling materials in primary teeth. ASDC J Dent Child. 2000 Mar-Apr;67(2):142-7, 83. No abstract available. PMID 10826052
- [Background] Amorim Lde F, Toledo OA, Estrela CR, Decurcio Dde A, Estrela C. Antimicrobial analysis of different root canal filling pastes used in pediatric dentistry by two experimental methods. Braz Dent J. 2006;17(4):317-22. doi: 10.1590/s0103-64402006000400010. PMID 17262146
- [Background] Mortazavi M, Mesbahi M. Comparison of zinc oxide and eugenol, and Vitapex for root canal treatment of necrotic primary teeth. Int J Paediatr Dent. 2004 Nov;14(6):417-24. doi: 10.1111/j.1365-263X.2004.00544.x. PMID 15525310
- [Result] Bonow MLM, Guedes-Pinto AC,Bammann LL. Antimicrobial activity of drugs used in pulp therapy of deciduous teeth. J EndodBraz, 1: 44-48, 1996
- [Result] Guedes-Pinto AC, De Paiva JG, Bozzola JR. [Endodontic treatment of deciduous teeth with pulp necrosis]. Rev Assoc Paul Cir Dent. 1981 May-Jun;35(3):240-4. No abstract available. Portuguese. PMID 6943625
- [Result] 14- Kramer PF, Faraco Junior IM, Feldens CA. Current status of pulp therapy in the Brazilian Universities - Pulpotomy and Pulpectomy Technique in deciduous teeth. J Bras Odontop e OdontolBebe, 3: 222-29, 2000.
- [Result] 16- Michel JA, Guedes-Pinto AC, AraújoVC. Estudo histopatológico da reação de subcutâneo de camundongos submetidos à ação da pasta Guedes-Pinto utilizada na terapia de dentes decíduos com polpa mortificada. RevFacOdontol São Paulo, 23: 65-72, 1980.
- [Result] Nurko C, Ranly DM, Garcia-Godoy F, Lakshmyya KN. Resorption of a calcium hydroxide/iodoform paste (Vitapex) in root canal therapy for primary teeth: a case report. Pediatr Dent. 2000 Nov-Dec;22(6):517-20. PMID 11132515